CLINICAL TRIAL: NCT06926036
Title: Micromanaging Human Sleep Physiology to Treat Sleep Apnea and Other Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Ken Paller, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FP00002577
Record Dates: First submitted 2025-03-05; First posted 2025-04-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Sleep Apnea Obstructive (OSA)
Keywords: sleep; sleep apnea obstructive (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental)
  Interventions: Behavioral: Wake training + TMR

INTERVENTIONS:
Behavioral: Wake training + TMR — In this within-participant design, all participants will undergo the same intervention of waking training and TMR.
  Waking training - waking training will associate an auditory cue with a specific learned behavioral response (a tongue protrusion and inhalation) during daily sessions for approximately one week, with home sleep monitoring.
  TMR - Targeted memory reactivation (TMR) refers to the process of playing learning-associated audio cues quietly during sleep in order to reactivate memories associated with the cue. After completion of waking training, TMR occurs in a laboratory setting, with PSG recording, during a single night.

SUMMARY:
This study will examine whether a combination of breathing training during wake and targeted reactivation of the training during sleep can induce breathing changes during sleep and subsequent cognitive benefits during wake.

Participants with obstructive sleep apnea (who have not yet been treated for sleep apnea) will be recruited. Participants will engage in breath training for one week in their own homes and to record their sleep at home using commercially available mobile devices and subsequently have their sleep monitored for one night of polysomnography recordings plus targeted reactivation in a laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handed, English-speaking adults, 18-60 years old who report normal hearing during sleep
2. Participants with suspected obstructive sleep apnea (OSA) (including those who have been diagnosed by a physician and those whose self-reported symptoms of OSA on the STOP-BANG questionnaire classify them as being "individuals with intermediate to high risk".
3. No report of any other sleep disorder besides OSA.
4. No report of any neurological or cardiometabolic diseases or disorders.
5. Not currently under active treatment for sleep apnea.
6. BMI ≤ 40.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | Day 1
  AHI indexes the severity of OSA on the night of the study.
Respiratory event duration | Day 1
  The duration of a hypopnea or apnea on the night of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ken A Paller, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No